CLINICAL TRIAL: NCT04249778
Title: Effect of Dapagliflozin at Discharge on Hospital Re-Admissions in Patients With Acutely Decompensated Heart Failure: A Randomized Controlled Study
Brief Title: Dapagliflozin at Discharge on Hospital Heart Failure Readmission
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00111588
Record Dates: First submitted 2020-01-14; First posted 2020-01-31 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Diabetes
Keywords: hospitalization; mortality; time of initiation of therapy; quality of life; cost-effectiveness; dapagliflozin; clinical trial; diabetes
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Patients admitted with exacerbation of chronic heart failure by clinical and radiologic features randomized to receive 10 mg of dapagliflozin, once daily for 26 weeks.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Patients admitted with exacerbation of chronic heart failure by clinical and radiologic features randomized to receive a placebo to match 10 mg of dapagliflozin, once daily for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin is a sodium-glucose cotransporter 2 (SGLT2) inhibitor indicated as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus. Participants will receive 10 mg/day of dapagliflozin, beginning at hospital discharge, for 26 weeks.
  Other Names: FARXIGA
  Arms: Dapagliflozin
Drug: Placebo — Participants will receive a placebo to match 10 mg/day of dapagliflozin, beginning at hospital discharge, for 26 weeks.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of dapagliflozin treatment in preventing hospital re-admissions, emergency room (ER) visits, urgent clinic visits, and death in patients with and without type 2 diabetes (T2D) after hospital admission for heart failure.

DETAILED DESCRIPTION:
The prevalence of both heart failure and type 2 diabetes (T2D) or prediabetes are reaching epidemic proportions globally and in the United States. More than 40% of patients with established heart failure (HF) have diabetes.

Dapagliflozin is a sodium-glucose cotransporter 2 inhibitor (SGLT2-i) indicated as an adjunct to diet and exercise to improve glycemic control in adults with T2D mellitus. Treatment with SGLT2-i has been shown to reduce both heart failure hospitalizations and mortality in patients with established heart disease. However, the time of initiation of SGLT2-i therapy has not been evaluated in patients with HF. This study will be the first trial to evaluate the safety and efficacy of dapagliflozin treatment in preventing hospital re-admissions, ER visits, urgent clinic visits, and death in patients with and without T2D after hospital admission for heart failure. In addition, the impact of treatment on HF symptoms quality of life, resource utilization, and cost-effectiveness of dapagliflozin versus placebo will be evaluated. The results of this study have great potential to impact and facilitate care and to change current clinical guidelines in the management of patients with heart failure.

Patients with and without diabetes who have acute decompensated heart failure (ADHF) will be randomized to take either dapagliflozin or placebo daily for 26 weeks, beginning at the time of discharge from from the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 90 years, with ADHF, and New York Heart Association (NYHA) class II, III, or IV symptoms discharged after hospital admission with a clinical diagnosis ADHF
2. Elevated natriuretic peptide tests measure levels of BNP (NT-pro-BNP) ≥300 pg/ml or B-type natriuretic peptide (BNP) ≥100 pg/ml on admission
3. Interpretable echocardiogram during hospital admission (or within 12 months prior to index hospitalization)
4. Blood glucose level <400 mg/dL without evidence of diabetic ketoacidosis (serum bicarbonate <18 milliequivalent (mEq)/L or positive serum or urinary ketones), in patients with T2D

Exclusion Criteria:

1. Age < 18 or > 90 years
2. Subjects with a history of type 1 diabetes
3. Treatment with thiazolidinediones (TZDs) or SGLT2-i during the past 3 months of admission
4. Recurrent episodes of severe hypoglycemia or hypoglycemic unawareness
5. History of recurrent HF admissions considered to be due to non-compliance (evaluated by the research staff for participation)
6. Patients with clinically significant hepatic disease (cirrhosis, jaundice, end-stage liver disease, portal hypertension) and elevated alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 3 times upper limit of normal
7. Patients with impaired renal function (GFR < 25 ml/min)
8. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
9. Patients on ventricular assist devices (VADs)
10. History of heart transplant or listed for heart transplant
11. History of cardiac surgery (within 90 days prior to enrollment) or planned cardiac interventions within the following 6 months, including percutaneous coronary intervention (PCI), ablation, cardiac resynchronization therapy (CRT) implantable cardioverter-defibrillator (ICD)
12. HF due to restrictive/infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, severe stenotic valvular diseases, hypertrophic cardiomyopathy, or congenital heart disease
13. History of SGLT2-i allergy
14. Systolic blood pressure < 100 mmHg
15. Uncontrolled hypertension, defined as a systolic blood pressure > 200 mmHg at randomization
16. Female subjects who are pregnant or breast-feeding at time of enrollment into the study
17. Females of childbearing potential who are not using adequate contraceptive methods
18. In hospice or expected life expectancy less than 6 months
19. Patients with diabetic foot infection, osteomyelitis and history of amputation of lower extremities within 6 months of admission
20. Patients anticipated to undergo major surgical procedures during the following 6 months
21. Patients with active hematuria, urinary tract infection (UTI), or history of frequent UTIs or genital mycotic infections
22. Uncontrolled atrial fibrillation or atrial flutter with a resting heart rate >110bpm documented by ECG at randomization
23. Any condition that in the opinion of the investigator would contraindicate the assessment of distance walked in 6 minutes (6MWD)
24. Chronic pulmonary disease, i.e. with known forced expiratory volume in the first second (FEV1) <50% requiring home oxygen, or oral steroid therapy or current hospitalization for severe chronic obstructive pulmonary disease (COPD) thought to be a primary contributor to dyspnea, or significant chronic pulmonary disease in the Investigator's opinion, or primary pulmonary arterial hypertension
25. Patients with active history of bladder cancer
26. Patients with previous history of diabetic ketoacidosis, per American Diabetes Association (ADA) criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Tulane University, New Orleans, Louisiana
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results reported, will be available for sharing after de-identification, including text, tables, figures, and appendices.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 6 months after publication of results from this study and ending 5 years after publication.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal. Proposals should be directed to geumpie@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three sites in the USA: Emory University Hospital in Atlanta, Georgia, Tulane University in New Orleans, Louisiana, and Temple University in Philadelphia, Pennsylvania. Participant enrollment began July 29, 2020 and all follow-up assessments were completed by March 3, 2022.
Groups:
- Dapagliflozin: Patients admitted to the hospital with exacerbation of chronic heart failure by clinical and radiologic features randomized to receive 10 mg of dapagliflozin, once daily.
- Placebo: Patients admitted to the hospital with exacerbation of chronic heart failure by clinical and radiologic features randomized to receive a placebo to match 10 mg of dapagliflozin, once daily.
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started (Participants who were randomized to a study arm) | 50 | 55
Started Study Medication | 46 | 53
Attended Week 12 Visit | 16 | 19
Completed (Completed the Week 26 visit) | 15 | 12
Not Completed | 35 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 50 | 55 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 45 | 85
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.12 (13.47) | 55.49 (11.63) | 55.79 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 10 | 40
  Male | 20 | 45 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 48 | 55 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 42 | 80
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 55 | 105
Diabetes Status [Count of Participants; unit: Participants]
  Diabetic (Type 2 Diabetes) | 21 | 17 | 38
  Non-diabetic | 26 | 31 | 57
  Pre-diabetic | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospital Admissions, Emergency Department Visits, Urgent Clinic Visits, and Death
Description: The number of participants meeting criteria for a composite of hospital admissions, emergency department visits, urgent clinic visits for heart failure and death after admission with acute decompensated heart failure (ADHF) was determined.
Time Frame: Up to 26 weeks
Population: This analysis includes participants who started the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
Participants | 0 | 3

2. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Score
Description: The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
score on a scale
  Baseline | 55.72 (23.23) | 50.71 (25.10)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 62.40 (37.52) | 66.95 (36.93)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 83.36 (13.51) | 80.38 (17.46)

3. Secondary Outcome: Chronic Heart Failure Questionnaire - Self-Administered Standardized Format (CHQ-SAS) Score
Description: Chronic Heart Failure Questionnaire - Self-Administered Standardized Format (CHQ-SAS) assesses patients' perception of their heart failure and measures the impact of heart failure symptoms. The CHQ-SAS contains 16 standardized questions that assess dyspnea during daily activities, fatigue and emotional function. Items are rated on a 7-point Likert scale ranging from 1 to 7. The total score is the mean of the item scores and higher scores indicate better quality of life.
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
score on a scale
  Baseline | 4.04 (1.51) | 4.07 (1.31)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 5.25 (1.05) | 5.34 (1.14)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 5.27 (0.93) | 5.27 (1.17)

4. Secondary Outcome: N-terminal (NT)-Pro Hormone BNP (NT-proBNP) Levels
Description: The heart failure, disease-specific biomarker N-terminal (NT)-pro hormone BNP (NT-proBNP) is a non-active prohormone. Levels increase when heart failure develops or gets worse and levels reduce when heart failure is stable.
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
picograms per milliliter (pg/mL)
  Baseline | 1947.38 (2641.03) | 1469.86 (1713.87)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 589.25 (391.37) | 1083.00 (1554.99)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 674.50 (388.71) | 730.00 (541.06)

5. Secondary Outcome: 6-Minute Walk Distance (6MWD)
Description: The 6-Minute Walk Distance (6MWD) test measures the distance, in meters, that a patient can quickly walk on a flat, hard surface in a period of 6 minutes
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants who started the study drug and who were physically able to partake in this assessment at the indicated study visits.
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 29 | 28
meters (m)
  Baseline | 893.42 (394.61) | 1109.05 (1271.43)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 1185.76 (321.27) | 1548.23 (1807.13)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 995.23 (414.59) | 1123.19 (379.64)

6. Secondary Outcome: Hemoglobin A1C (HbA1c) Level
Description: HbA1c was quantified by blood test, in participants with type 2 diabetes (T2D). Higher percentages of glycated hemoglobin on red blood cells (RBCs) indicate higher blood glucose levels in the previous three months. A normal HbA1c level is below 5.7 percent.
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants with type 2 diabetes who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: percent of RBCs with glycated hemoglobin
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 21 | 17
percent of RBCs with glycated hemoglobin
  Baseline | 9.41 (2.33) | 8.98 (1.91)
  Week 12: number analyzed (Participants) | 10 | 9
  Week 12 | 8.62 (2.12) | 8.47 (2.88)
  Week 26: number analyzed (Participants) | 6 | 5
  Week 26 | 9.47 (2.84) | 7.84 (2.38)

7. Secondary Outcome: Weight
Description: Weight is measured in kilograms.
Time Frame: Baseline,Week 12, Week 26
Population: This analysis includes participants who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
kilograms
  Baseline | 101.21 (35.77) | 103.59 (27.77)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 95.93 (30.26) | 101.18 (20.53)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 98.06 (29.05) | 100.18 (18.55)

8. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure is measured in millimeters of mercury (mmHg). A normal systolic blood pressure level is less than 120 mmHg.
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
mmHg
  Baseline | 124.39 (14.51) | 125.36 (17.38)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 118.15 (21.57) | 124.31 (19.88)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 131.69 (21.76) | 136.79 (23.69)

9. Secondary Outcome: Left Atrial Diameter
Description: The normal range for left atrial diameter is 2.0 to 4.0 centimeters (cm). The left atrium increases in size with heart conditions.
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
centimeters
  Baseline | 4.47 (0.79) | 4.32 (0.75)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 4.55 (0.82) | 4.91 (0.43)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 4.30 (1.12) | 4.31 (0.72)

10. Secondary Outcome: Serum Magnesium
Description: Normal levels of serum magnesium are between 1.7 and 2.3 milligrams per deciliter (mg/dL).
Time Frame: Baseline, Week 12, Week 26
Population: This analysis includes participants who started the study drug and attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
mg/dL
  Baseline | 2.01 (0.27) | 1.92 (0.48)
  Week 12: number analyzed (Participants) | 16 | 19
  Week 12 | 2.11 (0.22) | 2.02 (0.23)
  Week 26: number analyzed (Participants) | 15 | 12
  Week 26 | 2.13 (0.17) | 1.98 (0.27)

11. Secondary Outcome: Number of Participants Dying From Cardiovascular Reasons
Description: The number of participants dying due to cardiovascular reasons was documented.
Time Frame: Up to Week 26
Population: This analysis includes participants who started the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Non-fatal Myocardial Infarction (MI)
Description: The number of participants with non-fatal myocardial infarction (MI) was documented.
Time Frame: Up to Week 26
Population: This analysis includes participants who started the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Stroke
Description: The number of participants experiencing a stroke was documented.
Time Frame: Up to Week 26
Population: This analysis includes participants who started the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
Participants | 1 | 0

14. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: The number of participants experiencing acute kidney injury was documented.
Time Frame: Up to Week 26
Population: This analysis includes participants who started the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 46 | 53
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time individuals gave consent to participate in the study and continued through the Week 26 study visit.
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/55
Serious Adverse Events (participants affected / at risk) | 3/50 | 5/55
Other Adverse Events (participants affected / at risk) | 4/50 | 2/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=50) | Placebo (N=55)
Hospital readmission due to heart failure exacerbation (Cardiac disorders) | 0 | 3
Hospital readmission due to fall/weakness (General disorders) | 0 | 1
Hospital readmission due to chronic obstructive pulmonary disease (COPD) exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hospital readmission due to pneumonia (Infections and infestations) | 1 | 0
Hospital readmission due to gastroparesis (Gastrointestinal disorders) | 1 | 0
Hospital readmission due to cerebrovascular accident (CVA) (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=50) | Placebo (N=55)
Yeast infection (Infections and infestations) | 1 | 0
Peeling dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 (1)
ICD Implant (Surgical and medical procedures) | 0 | 1 (1)
Elective mitral valve replacement (Surgical and medical procedures) | 1 (1) | 0
Gout arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0

LIMITATIONS AND CAVEATS:
This study occurred during the Coronavirus Disease 2019 (COVID-19) pandemic resulting in many participants lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT04249778/Prot_SAP_000.pdf